CLINICAL TRIAL: NCT05977699
Title: Salbutamol Reversal of Methacholine Induced Bronchoconstriction: Vibrating Mesh Nebulizer Versus Pressurized Metered Dose Inhaler
Brief Title: Reversibility of Methacholine Induced Bronchoconstriction
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BIO 3632
Record Dates: First submitted 2023-06-19; First posted 2023-08-04 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- salbutamol delivered via pressurized metered dose inhaler (Active Comparator): 200mcg of salbutamol will be delivered using a pressurized metered dose inhaler plus spacer
  Interventions: Drug: salbutamol pressurized metered dose inhaler
- placebo (Placebo Comparator): normal saline will be administered with a vibrating mesh nebulizer and 200mcg of placebo will be administered using a pressurized metered dose inhaler plus spacer
  Interventions: Other: placebo
- salbutamol delivered with vibrating mesh nebulizer (Experimental): 200microliters of salbutamol will be administered using a vibrating mesh nebulizer
  Interventions: Drug: salbutamol aqueous solution

INTERVENTIONS:
Drug: salbutamol aqueous solution — administration of 200microliters of salbutamol to reverse methacholine induced bronchoconstriction using a vibrating mesh nebulizer
  Arms: salbutamol delivered with vibrating mesh nebulizer
Drug: salbutamol pressurized metered dose inhaler — administration of 200microliters of salbutamol to reverse methacholine induced bronchoconstriction using a pressurized metered dose inhaler plus spacer
  Arms: salbutamol delivered via pressurized metered dose inhaler
Other: placebo — matching placebo delivered via pressurized metered dose inhaler plus spacer or normal saline via vibrating mesh nebulizer
  Arms: placebo

SUMMARY:
The study will compare salbutamol reversibility of methacholine induced bronchoconstriction between a pressurized metered dose inhaler with a spacer versus nebulizer administration using a vibrating mesh nebulizer.

ELIGIBILITY:
Inclusion Criteria:

* age (years) at least 18, male or female
* no confounding health issue (i.e. no health conditions, other than asthma, that would put the participant at risk or affect data integrity)
* baseline FEV1 ≥ 65% predicted (per Quanjer GLI 2012)
* methacholine PD20 ≤ 800mcg

Exclusion Criteria:

* respiratory infection within 4 weeks of Visit 1
* exposure to triggers of respiratory symptoms within 4 weeks of Visit 1
* currently pregnant or breastfeeding
* current smoker (cigarettes, vaping)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Lung function recovery | up to 60 minutes post salbutamol administration
  Maximal recovery in FEV1 and FVC (absolute volume and percent)

SECONDARY OUTCOMES:
Time to lung function recovery | 0-60 minutes
  Area under the curve from start of salbutamol administration to time at which maximal recovery occurs
Heart rate | 0-60 minutes
  change in pulse after salbutamol administration

CONTACTS AND LOCATIONS:
Overall Officials: Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Asthma Research Lab University of Saskatchewan Room 346 Ellis Hall, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No